CLINICAL TRIAL: NCT05553249
Title: Written Exposure Therapy for PTSD: A Pilot Study of a Virtually Delivered Group-Based Intervention
Brief Title: Written Exposure Therapy for PTSD in a Virtual, Group-based Format
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HS25632 (H2022:260)
Record Dates: First submitted 2022-09-12; First posted 2022-09-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Virtual, group-based Written Exposure Therapy

SUMMARY:
The purpose of this study is to examine whether Written Exposure Therapy (WET) can be effectively delivered virtually and in a group format for the treatment of Post-Traumatic Stress Disorder in a military and police population. The objective of this study is to assess treatment feasibility and acceptability, drop out rates, changes in severity of trauma-related symptoms and symptoms of depression, quality of life, and the need for further trauma-focused treatment (TFT) for the the delivery of WET as a virtual, group based intervention.

DETAILED DESCRIPTION:
This study will assess the efficacy and acceptability of WET being delivered virtually and in a group format for the treatment of PTSD through the Operational Stress Injury Clinic (OSIC) at Deer Lodge Centre.

WET is offered in small groups of 10 patients. This study will follow 8 iterations of the group for a potential total of 80 participants in this study. Each WET group session will be facilitated by two OSIC clinicians, at least one of whom will be a clinical psychologist. Each session, administered via the Zoom app for healthcare, will start with a brief check in, then instructions will be provided to the whole group. Each group will receive a total of 5 therapy sessions, each of which will last approximately 1.5hrs.

Prior to the first WET session, participants will be asked to complete three clinical measures: Patient Health Questionnaire- 9 (PHQ-9), PTSD Checklist for DSM-5 (PCL-5, weekly version), and Outcome Questionnaire-45 (OQ-45). Participants will be asked to complete the PCL-5 prior to each session. Participants will also complete a Treatment Acceptability/Adherence Scale prior to the start of the second session.

Following the final session of therapy, participants will be asked to complete the three clinical assessment questionnaires (PHQ-9, PCL-5, and OQ-45) at 1 week, 1 month, and 3 months post-treatment. A research assistant will also follow-up with each participant at the 3-month mark to ask whether they have sought or attended further psychological treatment since the end of the WET sessions.

ELIGIBILITY:
Inclusion Criteria:

* Referred for Written Exposure Therapy at the Occupational Stress Injury Clinic (OSIC) in Winnipeg
* Able to speak, read, and write in English
* Medication held at a stable dose for four weeks prior to beginning treatment and throughout the duration of treatment (if on a prescribed medication)

Exclusion Criteria:

* Current psychosis
* Presence of another psychiatric disorder that requires prioritization over treating PTSD
* Any cognitive, visual, or motor impairment that would prevent writing for 30 minutes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Actively serving and veteran members of the Canadian Armed Forces and RCMP, previously diagnosed by a psychologist or psychiatrist with PTSD or Other Specified Trauma and Stressor-Related Disorder (meeting PTSD Criterion A), who have been referred to the OSIC for psychological treatment of their trauma-related disorder.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Treatment acceptability | 5 weeks
  Acceptability of the treatment program based on responses to the Treatment Acceptability/Adherence Scale. Scores on this scale range from 10-70 with higher scores indicating greater acceptability.

SECONDARY OUTCOMES:
Attrition | 5 weeks
  Rate of participant attrition from the treatment program
Change in PTSD symptoms | 5 weeks
  Change in PTSD symptom severity based on the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). Scores on this scale range from 0-80 with higher scores indicating greater symptom severity.
Psychotherapy progress | 5 weeks
  Psychotherapy progress as measured by the Outcome Questionnaire 45 (OQ-45). A total score of all subscales ranges from 0 to 180, with higher scores indicating more severe distress and functional impairment.
Change in depression symptoms | 5 weeks
  Change in depression symptoms based on the Patient Health Questionnaire-9 (PHQ-9). Scores on this scale range from 0-27, with higher scores indication more severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Bodkyn, PhD CPsych, Principal Investigator — University of Manitoba
Locations (1):
- Deer Lodge Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No